CLINICAL TRIAL: NCT02048800
Title: Evaluation of Treosulfan Pharmacokinetics (PK) in Children Undergoing Allogeneic Haematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Treosulfan Pharmacokinetics in Children Undergoing Allogeneic HSCT
Acronym: TreoPK
Status: Completed | Type: Observational
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 10MI28
Record Dates: First submitted 2014-01-17; First posted 2014-01-29 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Allogeneic Haematopoietic Stem Cell Transplantation
Keywords: Treosulfan pharmacokinetics; Children; Any condition that requires an allogeneic HSCT
MeSH Terms: interventions — treosulfan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma will be stored for Treosulfan PK analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treosulfan PK: Children with indication to HSCT receiving Treosulfan
  Interventions: Drug: Treosulfan

INTERVENTIONS:
Drug: Treosulfan — Treosulfan will be administered over 3 days prior to HSCT at the following dose: 10 g/m2 (children aged < 3months) or 12 g/m2 (children aged 3/12 months) or 14 g/m2 (children aged > 12 months)

SUMMARY:
Every year around 70 children affected by cancer or life-threatening genetic diseases undergo haematopoietic cell transplantation (HCT) within the Blood and Marrow Transplant (BMT) unit at Great Ormond Street Hospital (GOSH).

One of the main goals of the BMT unit over the last decade has been to reduce the morbidity and mortality related to HCT, and the group has become a world-leader in pioneering less toxic transplants.

Fixed high doses of chemotherapy drugs are generally used to prepare children for HCT but several studies have shown a correlation between the concentration of these drugs achieved in the patient's blood, and the success or failure of the HCT procedure.

Recently a new drug, Treosulfan, has become available for use in patients undergoing HCT, and GOSH has pioneered its introduction in children undergoing HCT. With promising early results, Treosulfan has become the pre-HCT drug of choice, however, very little is currently known about how the drug is metabolised and cleared from the body, particularly in children.

The investigators therefore plan to investigate the pharmacokinetic (PK) profile of Treosulfan in children undergoing HCT at GOSH and define which parameters affect its metabolism and clearance, and what blood levels are associated with a favourable outcome (graft take without toxicity) or a poor result (graft rejection and/or toxicity).

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 28 days and ≤ 18 years old;
2. Karnofsky Performance Status ≥ 50 or Lansky Performance Status ≥ 30;
3. provide signed, written informed consent from parent or guardian;
4. be able to comply with study procedures and follow-up examinations;
5. have adequate organ function (as indicated by Table 1, page 27), within 14 days prior enrollment;
6. negative pregnancy test in post-pubertal female patients.

Exclusion Criteria:

1. patients aged < 28 days and > 18 years old;
2. patients with compromised organ function*;
3. patients with any other severe concurrent disease, which, in the judgment of the Investigator, would make the patient inappropriate for entry into this study;
4. known hypersensitivity to Treosulfan or Fludarabine;
5. pregnancy/lactation.

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children affected by malignant or non-malignant diseases with an indication to allogeneic HSCT.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2014-03; Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
1) Assess maximum concentration (Cmax) after Treosulfan infusion in children prior to allogeneic haematopoietic stem cell transplantation. | day -7 and day -5 pre HSCT
2) Assess half life after Treosulfan infusion in children prior to allogeneic haematopoietic stem cell transplantation. | Day -7 and day-5 pre HSCT
3) Assess the area under the curve (AUC) after Treosulfan infusion in children prior to allogeneic haematopoietic stem cell transplantation. | Day -7 and day -5 pre HSCT

SECONDARY OUTCOMES:
1) Assess interindividual and intraindividual variability of PK parameters in children of different age and weight; | day -7 and -5 pre HSCT
  To measure Treosulfan PK parameteres such as maximum concentration, area under the curve and half life after the first (day -7) and third (day -5) dose of Treosulfan and study if there is any significant intrapatient and interpatient variability of these results.
2) Assess the relationship between PK parameters and patient characteristics; | day -7 and -5 pre HSCT
  To study the relationship between treosulfan PK parameters such as area under the curve, maximum concentration and half life after the 1st and 3rd administration and pre-HSCT parameters such as renal function (creatinine, urea levels) and liver function (ALT, AST, GGT, bilirubin).
3) Assess the relationship between Treosulfan PK and regimen related toxicity (using the NCI toxicity criteria scoring system) and survival; | from day -7 pre HSCT to day +100 post HSCT
  The toxicity of the transplant will be recorded in the clinical notes and CRF forms using the NCI toxicity criteria (toxicity score for every organ/system, with a range from 1 to 5). This information will be correlated to Treosulfan PK criteria such as maximum concentration and area under the curve
4) Assess the relationship between Treosulfan PK and efficacy parameters, such as rate of engraftment and donor chimerism. | from day -7 pre HSCT to day + 360 post HSCT
  Donor engraftment in the peripheral blood (in different cell lineages: CD15+ cells and CD3+ cells) will be addressed regularly after HSCT and these results will be correlated with Treosulfan PK parameters such as area under the curve.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Chiesa, MD, Principal Investigator — Great Ormond Street Hospital, London, UK; Mary Slatter, MD, Principal Investigator — Great North Childrens Hospital, Newcastle upon Tyne, UK
Locations (2):
- United Kingdom (2):
  - Great Ormond Street Hospital for Children, London
  - Great North Childrens Hospital, Newcastle upon Tyne

REFERENCES:
- [Background] Slatter MA, Rao K, Amrolia P, Flood T, Abinun M, Hambleton S, Nademi Z, Goulden N, Davies G, Qasim W, Gaspar HB, Cant A, Gennery AR, Veys P. Treosulfan-based conditioning regimens for hematopoietic stem cell transplantation in children with primary immunodeficiency: United Kingdom experience. Blood. 2011 Apr 21;117(16):4367-75. doi: 10.1182/blood-2010-10-312082. Epub 2011 Feb 16. PMID 21325599